CLINICAL TRIAL: NCT07083843
Title: The Effect of Non-pharmacological (Exercise Home-based Method) Intervention on Psychological Distress of Patients Undergoing Hemodialysis at Al-Suwaiq Renal Dialysis Center
Brief Title: Exercise Effect on Psychological Distress of Patients Undergoing Hemodialysis at Al-Suwaiq Dialysis Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oman Ministry of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MoH/CSR/24/28651
Record Dates: First submitted 2025-07-05; First posted 2025-07-24 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-09

CONDITIONS: Exercise; Renal Dialysis; Anxiety; Depression
MeSH Terms: conditions — Motor Activity; Anxiety Disorders; Depression | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group received home based exercise. (Experimental): Received home based exercise as following:
  1. Exercise (such as walking or biking) for 5 to 10 minutes. once a day or a few times throughout the day.
  2. Slowly adding 3 to 5 minutes to the exercise session. And keep adding time up to 30 to 60 minutes in 1 session.
  3. Begin exercising 2 to 3 days a week on the days free of a dialysis treatment.
  4. Then increase exercise session 4 to 7 times.
  Interventions: Behavioral: Exercise
- Control group (Active Comparator): This group will receive the standard care as usual.
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Behavioral: Exercise — Intervention, will receive home based exercise multi times per week for 6 months
  Arms: Intervention group received home based exercise.
Other: Standard medical treatment — Control group will receive the usual standard care.
  Arms: Control group

SUMMARY:
The aim to investigate the level of psychological distress on patients undergoing hemodialysis at Al-Suwaiq Renal dialysis center as well as to explore the effectiveness of home-based exercise method in reducing such psychological distress, depression, and anxiety.

the main questions aims to answer,

1. Does hemodialysis patients have high level of psychological distress.
2. Does exercise has effect on reducing psychological distress on hemodialysis patients.

participants randomized into control and intervention group, intervention group received home based exercise for 6 month while control group not, to compare in reducing of psychological distress.

DETAILED DESCRIPTION:
Patients with kidney failure undergoing hemodialysis experience psychological distress.Several psychosocial stressors have an impact on patients undergoing hemodialysis as dialysis treatment imposes several lifestyle changes. These include the impact of disease and treatment, dietary and fluid restrictions, functional limitations, sexual dysfunction, future uncertainty and fear of death. Commonly associated psychosocial issues include depression and anxiety. Exercise interventions may mitigate this outcome, but their clinical role is unclear. Thus. this project aims to examine the effect of non- pharmacological intervention exercise, walking, in reducing psychological distress.

This is a two-phases study in which a cross-sectional study will be conducted to evaluate the level of psychological distress among (n=132) patient undergoing hemodialysis at Al- Suwaiq renal dialysis center. as second phase patients randomize into two groups, One group will receive the non- pharmacological intervention (exercise home based) while the other group will continue the regular treatment plan. After 6 months of follow-up, a post-assessment of the psychological symptoms of the interventional and the control groups, using the same tool designed by University of Michigan Depression Center. A face-to-face survey will be applied among selected patients. A paired t-test will be used to assess the expected improvement due to the intervention program by comparing the pre-post assessments of psychological distress level. This study is expected to provide an alternative method of treatment to help renal patients to cope with their treatment consequences.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Diagnosis of ESRD on dialysis at least for 3 years
* Stable (no recent exacerbation).
* Not having Diabetic feet.
* Walking without assistance.

Exclusion Criteria:

* Any acute or chronic condition that would limit the ability of the patient to participate in the study.
* Refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Suwaiq Renal Dialysis unit., Sohar, Batinah North, Oman

IPD SHARING:
Plan to Share IPD: No
Saving patients data, confidentiality.

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30456545/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35194215/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30759022/
- See also: Related Info — https://journalkhd.com/ojs/index.php/htechj/article/view/301
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38048651/
- See also: Related Info — https://www.muscatdaily.com/2021/06/27/2500-chronic-kidney-disease-patients-in-oman/
- See also: Related Info — https://www.purepsychmi.com/a-pure-psychiatry-depression-anxiety?gad_source=1&gad_campaignid=22739141518&gbraid=0AAAAABXRYnpN7MuxPAVeWTuBa_kwoAWta&gclid=CjwKCAjwsZPDBhBWEiwADuO6ywHPMQ0l_tlq5G-3vqDWj_g4g8p5GwdqNYYTAYLz374agW_PLK2k6xoC2qUQAvD_BwE

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. Adults ≥18 years of age
  2. Diagnosis of ESRD on dialysis at least for 3 years
  3. Stable (no recent exacerbation).
  4. Not having Diabetic feet.
  5. Walking without assistance.
Pre-assignment Details: We started with 54 who were fit with our inclusion criteria, during second phase of intervention, one from intervention group withdraw as he is went into transplantation operation, and one from control group passed away. this lead as to 52 participants.
Groups:
- Intervention group.: after randomized fit patient and and doing pre assessment of psychological distress this group, received a non-pharmacological exercise home based program that includes:
  1. Exercise (such as walking or biking) for 5 to 10 minutes. once a day or a few times throughout the day.
  2. Slowly adding 3 to 5 minutes to the exercise session. And keep adding time up to 30 to 60 minutes in 1 session.
  3. Begin exercising 2 to 3 days a week on the days free of a dialysis treatment.
  4. Then increase exercise session 4 to 7 times. the intervention has been followed for 6 months.
- Control group: Received standard care as usual.
Period: assessment/data collection period.
Arm/Group | Intervention group. | Control group
Started | 27 | 27
Completed (to collect consent form, and pre assessment of psychological distress from 30/08/24 to 30/10/24) | 27 | 27
Not Completed | 0 | 0
Period: Intervention period.
Arm/Group | Intervention group. | Control group
Started | 27 | 27
Completed (follow up intervention monthly for 6 months, started from 1/11/24 to 31/4/25.) | 26 | 26
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 1
Period: follow-up
Arm/Group | Intervention group. | Control group
Started | 26 | 26
Completed (collecting post psychological assessment and analysis data, from 1/5/25 to 1/7/25) | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Received the standard care.
- Total: Total of all reporting groups
Arm/Group | Intervention Group. | Control Group | Total
Number analyzed (Participants) | 26 | 26 | 52
Region of Enrollment [Count of Participants; unit: Participants]
  Oman | 26 | 26 | 52
Generalized anxiety disorder. [Mean (Standard Deviation); unit: score on a scale (GAD-7)] — Through using approved survey from depression center of Michigan university, all participants were assessed before and after the intervention to measures any significant effect, this questionnaire consists of 7 questions with a four-point response option. The scoring is as follows: Low to mild anxiety severity (1-9 points), Medium anxiety severity (10-14 points), and High anxiety severity (15-21 points).
  score on a scale (GAD-7) | 4.8 (4.030) | 6.69 (4.412) | 5.75 (4.29)
Depression Scale [Mean (Standard Deviation); unit: score on a scale (PHQ_9)] — Through using approved survey from depression center of Michigan university, all participants were assessed before and after the intervention to measures any significant effect, this depression questionnaire consists of 9 questions with a four-point response option. with the scoring: Low depression severity (1-9 points), Medium depression severity (10-14 points), and High depression severity (15-27 points).applied face to face interviewing
  score on a scale (PHQ_9) | 2.96 (1.871) | 8.00 (5.710) | 5.48 (4.68)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 19 | 42
  >=65 years | 3 | 7 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 14 | 12 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression Score (PHQ-9) From Baseline to 6 Months.
Description: Depression severity was assessed using the PHQ-9 questionnaire ( patient health questionnaire-9), which consists of 9 questions rated on 4- points Likert scale from 0 (not at all)to 3 (nearly every day). the total score ranges from 0 to 27, with higher scores indicating more severe depression,
  Depression Severity levels :
  Low depression severity (1-9 points) Medium depression severity (10-14 points) and High depression severity (15-27 points). The outcome measure represents the change in PHQ-9 from baseline (pre- intervention) to 6 months post-intervention.
  The change in depression score was calculated by subtracting the score at 6 months from the score at baseline. this calculation was performed for both the intervention and control groups to evaluate the effectiveness of the exercise- based intervention.
Time Frame: Baseline (prior to intervention.) and 6 months after intervention.
Measure: Mean (Standard Deviation); unit: Unit on a scale.
Groups:
- control group: this group received standard care as usual.
Arm/Group | Intervention group. | control group
Number analyzed (Participants) | 26 | 26
Unit on a scale. | 2.96 (1.871) | 8.00 (5.710)
Statistical Analysis 1: Comparison: Intervention group. vs control group; Data was analyzed using SPSS v22.0., Descriptive statistics will summarize baseline variables. Paired t-test will assess pre- vs. post - intervention scores within groups, and between-group differences will be compared, the null hypothesis states there is no difference between intervention and control groups. A two-tailed P< 0.05 will be considered statistically significant; Test type: Superiority; p = 0.05, paired sample T-test; Degree of freedom = 25; Mean Difference (Final Values) = 4.115, 95% CI 2-sided [2.87 to 5.36], Standard Deviation 2.800

2. Primary Outcome: Change in Anxiety Score (GAD-7) From Baseline to 6 Months.
Description: Anxiety severity was assessed using the GAD-7 tool (General Anxiety disorder-7), which consists of 7 questions rated on 4- points Likert scale from 0 (not at all)to 3 (nearly every day). the total score ranges from 0 to 21, with higher scores indicating more severe anxiety,
  Anxiety Severity levels :
  Low Anxiety severity (1-9 points) Medium Anxiety severity (10-14 points) and High Anxiety severity (15-21 points). The outcome measrues represents the change in GAD_7 scores from baseline (pre-intervention) to 6 months post- intervention.
  The change in Anxiety score was calculated by subtracting the score at 6 months from the score at baseline. this calculation was performed for both the intervention and control groups to evaluate the effectiveness of the exercise- based intervention.
Time Frame: Baseline (prior to intervention.) and 6 months after intervention.
Measure: Mean (Standard Deviation); unit: Unit on a scale.
Arm/Group | Intervention group. | control group
Number analyzed (Participants) | 26 | 26
Unit on a scale. | 4.80 (4.030) [4.030 to 2.800] | 6.69 (4.412) [4.412 to 0.865]
Statistical Analysis 1: Comparison: Intervention group. vs control group; data were processed and analyzed using the SPSS software, version 22.0. The descriptive statistics were calculated, including frequencies and percentages for categorical data, and means and standard deviations for numerical variables. A paired t-test was used to assess the change in the psychological level before and after the intervention program. All hypothesis testing was done at the 5% level of significance; Test type: Superiority — A superiority analysis was performed to compare depression and anxiety scores between the intervention and control groups; p = 0.05, paired sample T-test; degree of freedom= 25; Mean Difference (Final Values) = 2.192, 95% CI 2-sided [0.986 to 3.238], Standard Deviation 2.800

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 6 months
Description: no adverse events were observed or reported during the study period.
Arm/Group | Intervention group. | control group
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

LIMITATIONS AND CAVEATS:
The study has several limitations. The sample size was relatively small (n=52 for final analysis), which may affect the generalizability of the findings. Adherence to the home-based exercise regimen was self-reported, which may introduce reporting bias or variability in actual physical activity levels. Additionally, The study duration was six months, which may not be sufficient to assess long-term sustainability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT07083843/Prot_001.pdf
  • Statistical Analysis Plan (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT07083843/SAP_002.pdf
  • Informed Consent Form (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT07083843/ICF_000.pdf